CLINICAL TRIAL: NCT05608863
Title: He-move-philia, a Combined Lifestyle Intervention Program for Patients With Hemophilia and Other Bleeding Disorders
Brief Title: He-move-philia, Lifestyle Intervention for Patients With Hemophilia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEMSTOL75
Record Dates: First submitted 2022-10-26; First posted 2022-11-08 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined intervention (Active Comparator): The Combined Lifestyle Intervention Program consists of a total of 7 individual coaching sessions and 16 group sessions in a 2 year program. The individual coaching sessions will be done in a virtual setting
  Interventions: Other: Lifestyle - group sessions
- individual intervention (Active Comparator): The Individual Intervention consists of a total of 7 individual coaching sessions in a 2 year program and additional written information. These will be done in a virtual setting
  Interventions: Other: Lifestyle - individual coaching

INTERVENTIONS:
Other: Lifestyle - group sessions — The Combined Lifestyle Intervention Program consists of a total of 7 individual coaching sessions and 16 group sessions in a 2 year program. The individual coaching sessions will be done in a virtual setting.
  Arms: Combined intervention
Other: Lifestyle - individual coaching — The Individual Intervention consists of a total of 7 individual coaching sessions in a 2 year program and additional written information. These will be done in a virtual setting.
  Arms: individual intervention

SUMMARY:
The main objectives are reduction of body weight, BMI and abdominal circumference. Secondary objectives are reduction of bleeds and units coagulation factor concentrate used, blood-pressure, cholesterol spectrum, glucose and improvement of physical activity and dietary habits. one group of patients will receive a combined lifestyle intervention program with individual sessions and group sessions lasting for 2 years, the other group of patients will receive individual sessions only and will be given the same information as given in the group sessions, but on paper.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity is increasing in patients with hemophilia and other bleeding disorders. In these patients physical activity is often difficult due to arthropathy as a result of intra-articular bleeding in the past, with decreased joint movement and pain and the fear of new bleeds. This enhances weight gain, increases pressure on joints, leading to more bleeds and more arthropathy. In the long term overweight and obesity increases risk of cardiovascular diseases, with the concomitant need for anticoagulant therapy, which further enhances the bleeding risk in these patients. The aim of this exploratory study is to compare the effect of a lifestyle intervention program consisting of combined individual coaching and group sessions (CLI) with a lifestyle intervention program with individual coaching only (II).The program is especially designed for patients with a bleeding disorder. The investigators hypothesize that body weight, BMI, abdominal circumference, bleeds and units coagulation factor concentrate, as these are dosed on body weight, will decrease in both groups, but more in the CLI with group sessions.

ELIGIBILITY:
Inclusion criteria

* Diagnosed with hemophilia A, B, FVII deficiency, fibrinogen deficiency, von Willebrand Disease or other bleeding disorder preferably requiring coagulation products for prophylaxis or on demand in case of bleeding
* ≥ 18 years of age
* BMI ≥ 30 kg/m2
* Motivated to change their lifestyle
* Being able to speak, read and understand the Dutch language

Exclusion criteria

* Health care insurance with CZ or ONVZ as these health insurances have no contract with Profitt Lifestylecoaching.
* A contraindication or inability for physical activity as judged by the treating hemophilia physician
* Participation in another research trial
* Unable to understand the written information
* Unable to sign the informed consent
* Unwilling to randomize to the combined or individual intervention group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
kg | 36 months
  The main study parameter is body weight in kg.

SECONDARY OUTCOMES:
Abdominal circumference (cm) | 36 months
Number of spontaneous bleeds | 36 months
Number of induced bleeds | 36 months
Units coagulation factor concentrate used/year (IU) | 36 months
Blood-pressurre (mm Hg) | 36 months
Cholesterol spectrum | 36 months
  including: total cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol (mmol/l), all in non-fasting state
Glucose (mmol/l) | 36 months
  in non-fasting state
Haemophilia activities of daily life (HAL) | 36 months
  Total score
Shortened Fat List | 36 months
  Total score

OTHER OUTCOMES:
BREQ-3 questionnaire | Baseline (week 0)
Regulation of Eating Behaviour Scale (REBS) | Baseline (week 0)
Patient satisfaction with the program will be measured using some questions | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Britta AP Laros - van Gorkom, MD, PhD, BSc, Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No